

## Statistical Analysis Plan

Study Code

PT003018 / FLUI-2015-139

Edition Number

1

Date

27 February 2017

A Randomized, Double-Blind, Two Treatment, Two Period, Chronic Dosing (2 Weeks), Cross-Over, Single-Center Study to Evaluate the Effects of PT003 and Placebo MDI on Specific Image Based Airway Volumes and Resistance in Subjects With Moderate to Severe COPD.

A Randomized, Double-Blind, Two Treatment, Two Period, Chronic Dosing (2 Weeks), Cross-Over, Single-Center Study to Evaluate the Effects of PT003 and Placebo MDI on Specific Image Based Airway Volumes and Resistance in Subjects With Moderate to Severe COPD

Study Statistician

A Randomized, Double-Blind, Two Treatment, Two Period, Chronic Dosing (2 Weeks), Cross-Over, Single-Center Study to Evaluate the Effects of PT003 and Placebo MDI on Specific Image Based Airway Volumes and Resistance in Subjects With Moderate to Severe COPD

Global Product Statistician

# **TABLE OF CONTENTS**

# **PAGE**

| | TITLE PAGE1 |
|---|---|
| | SIGNATURE OF STUDY STATISTICIAN2 |
| | SIGNATURE OF GLOBAL PRODUCT STATISTICIAN3 |
| | TABLE OF CONTENTS4 |
| | LIST OF ABBREVIATIONS6 |
| | AMENDMENT HISTORY8 |
| 1. | STUDY DETAILS9 |
| 1.1<br>1.1.1<br>1.1.2<br>1.1.3 | Study objectives9Primary objectives9Secondary objectives9Safety Objective9 |
| 1.2 | Study design9 |
| 1.3 | Number of subjects |
| 2. | ANALYSIS SETS11 |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4 | Definition of analysis sets |
| 2.2 | Violations and deviations |
| 3. | PRIMARY AND SECONDARY VARIABLES13 |
| 3.1<br>3.1.1<br>3.1.2<br>3.1.3<br>3.1.4<br>3.1.4.1<br>3.1.4.2<br>3.1.4.3 | Efficacy Endpoints13Definition of baselines13Treatment periods and visit windows13Primary Efficacy Endpoints13Secondary Efficacy Endpoints15FRI Parameters15Spirometry Parameters15Body Plethysmography Parameters16 |
| 3.1.4.3 | Other Efficacy Endpoints |
| 3.1.5.1<br>3.1.5.2 | FRI Parameters |
| 3.1.5.3 | Body Plethysmography Parameters |

| 3.2 | Safety Endpoints | 18 |
|---|---|---|
| 3.3 | Handling of missing data | 19 |
| 4. | ANALYSIS METHODS | 19 |
| 4.1<br>4.1.1 | General principles | |
| 4.1.2 | Hypothesis testing<br>Control of Type I error | 20 |
| 4.1.3 | Software | 20 |
| 4.2 | Analysis methods | 20 |
| 4.2.1 | Disposition, demographics and baseline characteristics | |
| 4.2.2 | Concomitant medications | 21 |
| 4.2.3 | Exposure and compliance | 21 |
| 4.2.4 | Analysis of FRI data | 21 |
| 4.2.5 | Spirometry / Body Plethysmography data | |
| 4.2.6 | Assumptions Checks and Removal of Outliers in Sensitivity Analyses | |
| 4.2.7 | Exploratory analyses | |
| 4.2.8 | Safety data | |
| 5. | INTERIM ANALYSES (NOT APPLICABLE) | 24 |
| 6. | CHANGES OF ANALYSIS FROM PROTOCOL | 24 |
| 7. | REFERENCES | 24 |
| 8. | APPENDIX | 25 |

# LIST OF ABBREVIATIONS

| AE Adverse Event ATC Anatomic Therapeutic Class ATS American Thoracic Society BID Bis In Die, twice daily CFD Computational Fluid Dynamics COPD Chronic Obstructive Pulmonary Disease CSR Clinical Study Report CT Computed Tomography ECG Electrocardiograms eCRF electronic Case Report Form ERS European Respiratory Society FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV1 Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
|---|
| ATS American Thoracic Society BID Bis In Die, twice daily CFD Computational Fluid Dynamics COPD Chronic Obstructive Pulmonary Disease CSR Clinical Study Report CT Computed Tomography ECG Electrocardiograms eCRF electronic Case Report Form ERS European Respiratory Society FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV1 Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| BID Bis In Die, twice daily CFD Computational Fluid Dynamics COPD Chronic Obstructive Pulmonary Disease CSR Clinical Study Report CT Computed Tomography ECG Electrocardiograms eCRF electronic Case Report Form ERS European Respiratory Society FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV1 Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| CFD Computational Fluid Dynamics COPD Chronic Obstructive Pulmonary Disease CSR Clinical Study Report CT Computed Tomography ECG Electrocardiograms eCRF electronic Case Report Form ERS European Respiratory Society FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV1 Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| COPD Chronic Obstructive Pulmonary Disease CSR Clinical Study Report CT Computed Tomography ECG Electrocardiograms eCRF electronic Case Report Form ERS European Respiratory Society FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV <sub>1</sub> Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| CSR Clinical Study Report CT Computed Tomography ECG Electrocardiograms eCRF electronic Case Report Form ERS European Respiratory Society FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV <sub>1</sub> Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| CT Computed Tomography ECG Electrocardiograms eCRF electronic Case Report Form ERS European Respiratory Society FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV <sub>1</sub> Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| ECG Electrocardiograms eCRF electronic Case Report Form ERS European Respiratory Society FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV <sub>1</sub> Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| eCRF electronic Case Report Form ERS European Respiratory Society FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV <sub>1</sub> Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| ERS European Respiratory Society FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV <sub>1</sub> Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| FEF25-75 Forced Expiratory Flow between 25% to 75% of FVC FEV <sub>1</sub> Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| FEV <sub>1</sub> Forced Expiratory Volume In 1 Second FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| FRC Functional Residual Capacity FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| FRI Functional Respiratory Imaging FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| FVC Forced Vital Capacity GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| GFF Glycopyrronium and Formoterol Fumarate GOLD Global initiative for chronic Obstructive Lung Disease |
| GOLD Global initiative for chronic Obstructive Lung Disease |
| 8 |
| HFA Hydrofluoroalkane |
| IC Inspiratory Capacity |
| IPD Important Protocol Deviation |
| iRaw Image based Airway Resistance |
| ITT Intent-To-Treat |
| iVaw Image based Airway Volume |
| iVlobe Image based Lobar Volume |
| LUL Left Upper Lobe |
| LL Lower Lobe |
| LLL Left Lower Lobe |
| MDI Metered Dose Inhaler |
| mITT Modified Intent-To-Treat |
| PFT Pulmonary Function Test |
| Raw Airway Resistance |
| RLL Right Lower Lobe |
| RML Right Middle Lobe |
| RUL Right Upper Lobe |

| Abbreviation or special term | Explanation |
|------------------------------|-------------------------------------------|
| RV | Residual Volume |
| sGaw | Specific Airway Conductance |
| siRaw | Specific Image based Airway Resistance |
| siVaw | Specific Image based Airway Volume |
| sRaw | Specific Airway Resistance |
| TEAE | Treatment Emergent Adverse Event |
| TLC | Total Lung Capacity |
| TP | Treatment Period |
| UA | Upper Airway |
| UL | Upper Lobe |
| WHO-DD | World Health Organization Drug Dictionary |

# AMENDMENT HISTORY

| Date | Brief description of change |
|------|-----------------------------|
| | N/A |

#### 1. STUDY DETAILS

# 1.1 Study objectives

# 1.1.1 Primary objectives

 To assess the effect of treatment with Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI), twice daily (BID) compared with Placebo MDI on specific image-based airway volumes and resistance in subjects with moderate to severe chronic obstructive pulmonary disease (COPD) following chronic dosing after approximately two weeks treatment.

## 1.1.2 Secondary objectives

- To compare the effects of GFF MDI on various Functional Respiratory Imaging (FRI) parameters.
- To compare the effects of GFF MDI and Placebo MDI on pulmonary function test (PFT) parameters.

## 1.1.3 Safety Objective

To assess the safety of GFF MDI in subjects with moderate to severe COPD based on adverse events (AEs), and any clinically relevant findings from vital sign measurements, electrocardiograms (ECGs), physical examination findings and clinical laboratory evaluations.

# 1.2 Study design

This is a single center, double-blind, two treatment, two period, full cross-over, chronic dosing (2 weeks) study to assess the effects of GFF MDI (14.4/9.6 µg BID) compared with Placebo MDI BID on specific image-based airway volumes and resistance in subjects with moderate to severe COPD.

Approximately 20 patients will be randomised to one of two sequences (GFF MDI followed by Placebo MDI or Placebo MDI followed by GFF MDI)

The sensitivity of the study increases with the crossover design where each subject acts as his/her own control. In this study the calculation of airway dimension parameters between the active compound and the placebo will be compared within the same subject after the administration of both the active compound as well as the placebo.

This single-center study will be conducted at one site in Belgium, with the site contributing approximately 20 randomized subjects with moderate to severe COPD.

## **Study Duration:**

Each subject will receive in total study treatment for approximately 4 weeks in two separate treatment periods of two weeks. Between the Treatment Periods there will be a washout

period of 5-21 days. The entire study is scheduled to take approximately 13 weeks for each individual subject.

# Study design chart



# Computed Tomography (CT)-scans during study:

On Day 1 of each Treatment Period [Visit 2 and Visit 4] a baseline measurement inspiratory scan (total lung capacity [TLC] scan) and expiratory scan (functional residual capacity [FRC] scan) will be conducted. During Visit 2 an additional scan of the upper airway (UA) will be taken. Post dose measurement inspiratory scan (total lung capacity [TLC] scan) will be taken after approximately 2 weeks of treatment with either GFF MDI or Placebo MDI on Day 15 (± 5 days) (Visit 3 and Visit 5). Post dose activities should be started 1 hour after dosing on Visit 3 and Visit 5 and should be concluded within 2.5 hours after dosing.

# 1.3 Number of subjects

Approximately 20 subjects with moderate to severe COPD will be randomized into the study

In a double blind cross over study where 10 COPD Global Initiative for Chronic Obstructive Lung Disease (GOLD) III subjects received a budesonide/formoterol combination, FRI was able to quantify the effects of the active compound relative to placebo. A sample size calculation (power goal 90%, alpha 0.05) revealed that in order to have a well-powered study with change in imaging based airway volume as primary outcome parameter, a total of 7 subjects would be required (De Backer, 2012). This is based upon powering for a difference of around 1 mL in iVaw and assuming a standard deviation of within subject differences of around 0.6 mL. Similarly, 17 subjects would be required for the image based airway resistance. If the significance level for the volume is set to 0.025 by the Hochberg's step-up procedure, 8 subjects would be required. It can be assumed that a good power will be obtained when including 20 subjects.

## 2. ANALYSIS SETS

# 2.1 Definition of analysis sets

The following analysis populations are defined in this study:

# 2.1.1 Intent-To-Treat (ITT) population

The ITT Population is defined as all subjects who are randomized to treatment. Data are analysed by randomized treatment regardless of the treatment actually received.

## 2.1.2 Modified Intent-To-Treat (mITT) population

The modified Intent-to-Treat (mITT Population) is a subset of the ITT population including subjects who received treatment and have post treatment efficacy data from both Treatment Periods. Data judged to be impacted by important protocol deviations will be determined prior to unblinding and excluded. Statistical tabulations and analyses will be by randomized treatment, but data obtained after subjects receive an incorrect treatment will be excluded from the affected periods.

## 2.1.3 Safety population

The Safety Population is defined as all subjects who are randomized to treatment and receive at least one dose of the study treatment. Statistical analyses and tabulations will be by the treatment actually received.

# 2.1.4 Population for analyses

Analyses will be performed as follows:

Demographics will be summarized for the ITT population. Extent of exposure will be summarized for the Safety Population. The Safety Population will be used to summarize safety data.

Efficacy analyses will be performed for the ITT Population. If the mITT Population differs from the ITT Population it will be used to conduct sensitivity analyses for the co-primary endpoints.

### 2.2 Violations and deviations

Only Important Protocol Deviations (IPDs) will be listed or tabulated. These are defined as those protocol deviations that may significantly affect the completeness, accuracy, and/or reliability of the study data or that may significantly affect a patient's rights, safety, or well-being. These will be identified based upon blinded data, before database lock.

The following will be considered important protocol deviations:

- Patient randomized despite not meeting key inclusion criteria, including:
  - O Patients not meeting COPD diagnosis (as defined by ATS/ERS) and severity criteria (FEV<sub>1</sub>/FVC ratio of <0.70 and post-bronchodilator FEV<sub>1</sub> >30% and <80% of predicted normal) as per inclusion criteria 5 and 7.
  - O Patients meeting exclusion criteria for other respiratory disease as per exclusion criteria 4, including diagnoses of asthma.
- Patient received incorrect study drug
- Prohibited concomitant COPD medication taken during the study, defined as the classes of medications listed in table 5-1 of the protocol, received after visit 2, other than those provided by the sponsor.
- Developed discontinuation criteria but not withdrawn from study or discontinued investigational product

#### Randomization errors

If a subject is given a treatment pack for a different patient or is randomized out of chronological order, he will be included in the statistical analysis. If a subject would receive the same treatment twice, this will be considered an important protocol deviation and sensitivity analyses will be conducted using the mITT population.

# 3. PRIMARY AND SECONDARY VARIABLES

# 3.1 Efficacy Endpoints

#### 3.1.1 Definition of baselines

Efficacy baseline assessments are taken pre-dose at Day 1 of each Treatment Period (TP) (Visits 2 and 4). The mean of the available pre-dose assessments across both of these visits will be taken as the subject-average baseline. The mean of the available pre-dose assessments at each of Visit 2 and Visit 4 respectively will be taken as the period-dependent baseline for that respective TP.

For spirometry and plethysmography endpoints the subject-average baseline will be used. That is the mean of all available pre-dose values conducted at Day 1 of each TP will be used to establish baseline. For spirometry the mean of the pre-dose -60 and -30 minute values at Visit 2 and Visit 4 will be averaged. In patients missing either of these assessments the single value from that visit will be used. Baselines for plethysmography endpoints will be based upon the -30 minute assessments.

For FRI parameters subject-average baselines will be derived for each patient as the mean of the baselines across all lobes and periods. Similarly subject-by-period average baselines will be derived across lobes at the subject by period level. These will be used as covariates in sensitivity analyses, but the primary analysis will be conducted on absolute values at Day 15 without using baseline covariates.

#### 3.1.2 Treatment periods and visit windows

There will be two treatment periods in this study. The first day on which a study treatment is received is Treatment Day 1 (for that study treatment and period). Treatment day is numbered sequentially thereafter until washout is begun or a subsequent study treatment is received. Each treatment period is intended to last until Day15.

No study time windows will be derived for the reporting of data. Data will be reported according to the protocol-scheduled day. Efficacy data obtained during unscheduled visits after Day 1 will be allocated to Day 15 within the same treatment period if the Day 15 visit is missing. For analysis of spirometry data by time point, if multiple values are collected the last available assessment will be used for a given nominal time point.

## 3.1.3 Primary Efficacy Endpoints

# **FRI Parameters:**

The co-primary endpoints of this study are as follows:

• Specific Image based airway volume (siVaw): Absolute value in Airway Volume (iVaw) relative to the lobar volume at Day 15.

• Specific Image based airway resistance (siRaw): Absolute value in Airway Resistance relative to the lobar volume at Day 15.

For FRI parameters data is generated within each of the five lobes of the lung (right upper lobe, right middle lobe, right lower lobe, left upper lobe and left lower lobe). Only the trimmed iVaw values will be taken for the derivation of these parameters.

For FRI parameters, only data generated from the scans taken at TLC level will be used for statistical analyses, but data generated at FRC will also be listed and will be summarised for selected parameters.

Visible airway generations can be different in the pre-dose CT and the post-dose CT scans. For the primary outcome, the airways are trimmed until the same length for both visits. We thus only asses the generations of airways that are visible in the scans of both study visit days. This allows us to view the pure bronchodilation of the airways.

The values of siVaw and siRaw are derived from iVaw and iRaw by dividing iVaw by the image based lobe volume (iVlobe) for siVaw and by multiplying iRaw by iVlobe for siRaw. See the definitions of iVaw, iRaw and iVlobe below. On a lobar scale (RUL: right upper lobe, RML: right middle lobe, RLL: right lower lobe, LUL: left upper lobe, LLL: left lower lobe), these calculations are:

- siVaw LLL = iVaw LLL / iVlobe LLL
- siVaw LUL = iVaw LUL / iVlobe LUL
- siVaw RML = iVaw RML / iVlobe RML
- siVaw RUL = iVaw RUL / iVlobe RUL
- siVaw RLL = iVaw RLL / iVlobe RLL
- siRaw LLL = iRaw LLL \* iVlobe LLL
- siRaw LUL = iRaw LUL \* iVlobe LUL
- siRaw RML = iRaw RML \* iVlobe RML
- siRaw RUL = iRaw RUL \* iVlobe RUL
- siRaw RLL = iRaw RLL \* iVlobe RLL

Similarly, values can be derived for the Lower Lobe (LL) by first summing iVaw values for LLL and RLL or for the Upper Lobe (UL) by first summing iVaw values for the LUL, RML and RUL. Distal totals can be derived using all 5 lobes. For airflow and resistance parameters a result from the central region of the lung is also provided and this combined with the distal total gives an overall total. For deriving resistance totals, parallel sums of iRaw should be used, by summing the inverse of iRaw values and then inverting again.

For FRI parameters the values for each lobe, the lower lobe total, upper lobe total and overall total will be listed.

# 3.1.4 Secondary Efficacy Endpoints

#### 3.1.4.1 FRI Parameters

• Airway volume (iVaw): Absolute value at Day 15

In the CT scans, the airways can be segmented up to the point where no distinction can be made between the intraluminal and alveolar air. This is where the airway diameter is around 1-2 mm, typically around the 5th to 10th bifurcation, depending mainly on the disease state of the individual patient. From the resulting model, the central and distal airway volumes can be assessed at individual airways or in different regions.

The distal airway volume is defined as the segmented airway volume starting from the third bifurcation, that is from the 5 lung lobes without the central region. It is this distal region that will be used in the analyses in this study.

Visible airway generations can be different in the pre-dose CT and the post-dose CT scans. The iVaw measurements can be performed in two ways: 1) measure of all the generation visible at certain study visit day 2) only assess the generations of airways that are visible in the scans of both pre-dose CT and the post-dose CT scans. The first parameter is called untrimmed iVaw and gives us an idea of the bronchodilation and bronchial recruitment, while the second parameter, called trimmed iVaw, allows us to view the pure bronchodilation. Both iVaw parameters will be analysed.

• Airway resistance (iRaw): Absolute value at Day 15

The airway resistance (iRaw) is determined using Computational Fluid Dynamics (CFD). During the CFD calculations, the outflow to each lobe is adjusted iteratively for each patient to match the internal flow rate distributions obtained from the segmentation of the CT scans hence iRaw accounts for the patient specific internal airflow distribution which might be greatly altered by the lung disease. Hence, the airflow distribution in the CFD calculation reflects the airflow distribution as derived from the expansion of the lung lobes from FRC to TLC. The iRaw is defined as the total pressure drop over an airway, divided by the flow rate through that airway.

Visible airway generations can be different in the pre-dose CT and the post-dose CT scans. For iRaw, the airways are trimmed until the same length for both visits. We thus only asses the generations of airways that are visible in the scans of both study visit days.

#### 3.1.4.2 Spirometry Parameters

• Forced expiratory volume in one second (FEV<sub>1</sub>): Change from baseline to Day 15 in post-dose FEV<sub>1</sub>

The volume of air exhaled under forced conditions in the first second. Post-dose results will be used. Change from baseline is calculated relative to the subject-average baseline.

# 3.1.4.3 Body Plethysmography Parameters

• Functional residual capacity (FRC): Change from baseline to Day 15 in post-dose FRC

The volume in the lungs at the end-expiratory position. Change from baseline is calculated relative to the subject-average baseline.

# 3.1.5 Other Efficacy Endpoints

#### 3.1.5.1 FRI Parameters

The following parameters will be analysed formally using scans at TLC with the exception of the mass of deposited particles, Internal Airflow Distribution and Air Trapping, which will be summarised descriptively only.

• Image based Lobe volumes (iVlobe): Absolute value at Day 15

By identifying and grouping the voxels that represent the air in the lungs the lung volume (L) can be determined from the scans. During segmentation, identifying the fissure planes on the CT images and using these surfaces as cutting objects can separate lung lobes. This means that not only the total lung volume is determined, but also the volume of each lobe individually.

For each treatment, only scans at the TLC level are taken after the treatment. That means that analyses can only be performed on TLC lobar volumes but not for FRC. For the FRC level, only descriptive summary of baseline values will be presented.

The percent predicted image based lobe volume (based upon age, sex and height) will also be derived. This will be analysed similarly to iVlobe using scans at the TLC level and summarised at baseline using scans at the FRC level.

• Air trapping: Descriptive summary of baseline results

Air trapping is defined as all the intrapulmonary voxels with Hounsfield Units between -1024 and -850 using the expiratory scans at FRC. This parameter is given as percentage of iVlobe.

Air Trapping is only valid on FRC scans, so because there are no FRC scans after treatment, no analyses can be done, only descriptive summary of baselines values. The air trapping will also be derived for the upper lobes, lower lobes and total by summing data from relevant individual lobes.

Internal lobar airflow distribution: Descriptive summary of baseline results

By segmenting the lobes at FRC and TLC for each patient, the patient-specific airflow distribution can be established by assessing lobar volume expansion.

Internal Airflow Distribution requires both FRC and TLC scans, so because there are no FRC scans after treatment no analyses can be done. Only descriptive summary of baselines values will be produced.

Low attenuation or emphysema score: Absolute value at Day 15

Low attenuation score is defined as all the intrapulmonary voxels with Hounsfield Units between -1024 and -950 using the inspiratory scans at TLC. This parameter is given as percentage of iVlobe.

Blood vessel density or fibrosis score: Absolute value at Day 15

Blood vessel density can be determined through segmentation and three-dimensional reconstruction of the blood vessels. The segmentation is based on a Hounsfield unit (HU) threshold between -600 and 600 and is performed on the TLC scan. The blood vessel density can be considered a surrogate for perfusion. This parameter is given as percentage of iVlobe.

• Airway wall thickness: Absolute value at Day 15

The airway wall volume consists of all visible tissue in the CT scan that encompasses the airway wall. The airway wall volume can typically be described to the same generation level as the volume description of the airway lumen, this is where the airway diameter is around 1 - 2 mm. This parameter can also be given relative to the lobar volume and is then called specific airway wall volume (siVaww). Visible airway generations can be different in the pre-dose CT and the post-dose CT scans. For airway wall thickness, the airways are trimmed until the same length for both visits. We thus only asses the generations of airways that are visible in the scans of both study visit days.

• Mass of deposited particles per defined airway section: Descriptive summary of baseline results

Regional aerosol deposition is determined by simulating the flow in the patient specific geometries using patient specific boundary conditions by means of CFD. While solving the flow equations, simultaneously particles are released in the flow and the force mass balance of the individual particles is determined through additional discrete phase computations. When a calculated particle trajectory intersects with the airway wall, the particle is trapped in that location. This allows determining the regional concentration of inhaled aerosols and consequently the effective lung dose of inhaled medication. These are measured in the full airway tree.

Mass of deposited particles is a useful way to see the particle deposition in each region of the lung. Data from the baseline TLC scan will be summarised. Distal and peripheral data will be summed. Upper lobe and lower lobe totals will also be derived.

# 3.1.5.2 Spirometry Parameters

The change from baseline at Day 15 will be assessed for the following parameters. Change from baseline is calculated relative to the subject-average baseline.

- Forced vital capacity (FVC): the determination of the vital capacity from a maximally forced expiratory effort
- Tiffeneau index (FEV<sub>1</sub>/FVC ratio): the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration
- Forced expiratory flow 25%-75% (FEF25-75): forced expiratory flow at 25–75% of forced vital capacity
- Inspiratory capacity (IC): the amount of air that can be inhaled after the end of a normal expiration. The average of the available Day 15 post-dose assessments will be used.

# 3.1.5.3 Body Plethysmography Parameters

The change from baseline at Day 15 will be assessed for the following parameters. Change from baseline is calculated relative to the subject-average baseline.

- Residual volume (RV): the volume of air remaining in the lungs after a maximal exhalation
- TLC: the volume in the lungs at maximal inflation
- Airway resistance (Raw): the resistance of the respiratory tract to airflow during inspiration and expiration
- Specific airway resistance (sRaw): airway resistance corrected for differences in lung volume. Specific airway conductance (sGaw): derived as the mathematical inverse of airway resistance corrected for differences in lung volume

# 3.2 Safety Endpoints

The safety assessments include Adverse Events (AEs) and Serious Adverse Events (SAEs) during the study period.

AEs experienced by the subjects will be collected throughout the entire study and will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA).

Only treatment emergent adverse events from the time of randomization onwards will be summarised. AEs will be assigned to the treatment period in which they first occurred. AEs reported as starting during a Washout Period or follow-up period will be assigned to the last treatment received. If an AE has a missing or partial onset date, then unless the stop date of the AE indicates otherwise, this will be considered an on treatment event.

Clinically relevant findings from laboratory, ECG and vital sign parameters will be reported as adverse events. As such these assessments will not be further tabulated.

# 3.3 Handling of missing data

Data for FRI parameters will be generated across each lobe of the lung. For an individual there may be missing data within certain lobes if for example the subject is missing that lobe or no airways lead to the lobe (giving a volume of zero and infinite airway resistance). If fissures between lobes cannot be distinguished then only a combined estimate across multiple lobes may be produced. Such results from combined lobes will not be used in the analyses. This will be consistent for both periods. Such combined lobe results may however enable totals and sub-totals to be calculated for a patient if the lobes which are combined coincide with those required for relevant regions.

Data from all individually evaluable lobes will be used in the analysis to allow for the estimation of effects at the subject level across all lobes. For patients with lobes that cannot be distinguished the estimates for that lobe are not meaningful for the patient and so they will not contribute, but this will be the case for both periods. Where scans are not evaluable for a single assessment or period this data is assumed to be missing at random.

Where Day 15 assessments are missing data from unscheduled post-baseline assessments will be used in their place, if available. No further imputation for missing values is planned.

#### 4. ANALYSIS METHODS

The primary objective of this study is to assess the effect of treatment with GFF MDI, 14.4/9.6 µg ex actuator, BID relative to Placebo MDI BID on specific image based airway volumes and resistance in subjects with moderate to severe COPD.

# 4.1 General principles

# 4.1.1 Hypothesis testing

For the efficacy analyses, the null hypothesis for each pair-wise comparison will be that the mean GFF MDI treatment effect is equal to that of Placebo MDI; the alternative hypothesis is then that the GFF MDI treatment effect and that of Placebo MDI are not equal. P-values will thus be reported as two-sided. Statistical level of significance will be set to 0.05.

For the co-primary endpoints and other FRI parameters the effect is defined using the absolute value at Day 15 of each TP. For the spirometry and plethysmography parameters the effect is defined in terms of the change from baseline, given that these parameters are commonly reported in those terms.

The null (H0) and alternative (H1) hypotheses with  $\mu$  representing the mean are:

H0:  $\mu_{GFF} = \mu_{placebo}$ 

H1:  $\mu_{GFF} \neq \mu_{placebo}$ 

For each parameter in each group this null hypothesis will be tested. The different groups are:

- Primary efficacy endpoints: FRI
- Secondary efficacy endpoints: FRI; Spirometry and Body Plethysmography
- Other efficacy endpoints: FRI parameters (except the mass of deposited particles, internal airflow distribution and air trapping); Spirometry and Body Plethysmography

In order to gain extra insight into the mode of action of the product, additional exploratory analyses may be executed using (robust) linear regression or mixed-models if necessary and reported outside of the Clinical Study Report (CSR).

The Intent-to-Treat (ITT) Population will be considered the primary analysis population for efficacy.

Continuous efficacy variables will be summarized with descriptive statistics (the number of non-missing values, mean, standard deviation, median, minimum and maximum). Where data has been logarithmically transformed for analysis the summary statistics on the backtransformed data will include the geometric mean and the coefficient of variation (calculated as  $100x\sqrt{[exp(s^2)-1]}$ , where s is the standard deviation of the data on the log scale. Categorical variables will be summarized with frequency counts and percentages, by treatment.

Only data deemed to meet acceptability criteria, for example regarding the quality of spirometry procedures, will be listed and summarised.

## 4.1.2 Control of Type I error

For the primary efficacy endpoints, Hochberg's step-up procedure will be used as multiplicity adjustment. No correction will be performed for the secondary and the other efficacy endpoints.

#### 4.1.3 Software

All statistical analysis will be conducted using R version 3.0.2 or higher (The R Foundation for Statistical Computing, Vienna, Austria), SAS version 9.2 or higher, or other validated software as appropriate.

# 4.2 Analysis methods

#### 4.2.1 Disposition, demographics and baseline characteristics

Descriptive summaries of disposition, demographics and baseline characteristics will be produced. Disposition tables will summarise the number of patients who received each treatment, the number who completed 1 or 2 treatment periods and the number of early

discontinuations. The number of patients in each analysis set will be summarised along with any reasons for exclusion.

Demographics and baseline characteristics at screening will be summarised descriptively, including COPD disease duration and symptom severity scores. Baseline pre and post bronchodilator spirometry parameters and reversibility to Ventolin HFA will be summarised using descriptive statistics based upon the baseline assessments within each treatment period.

#### 4.2.2 Concomitant medications

Concomitant medications will be will be assigned a preferred term and an ATC (Anatomic Therapeutic Class) term using the latest version of the World Health Organization Drug Dictionary (WHO-DD) available. Medications will be summarised according to whether they are COPD related or non-COPD related. Summaries will be presented for those medications started prior to the beginning of study treatment, those started during a treatment period and those started during the washout period.

## 4.2.3 Exposure and compliance

The number of days of exposure to each treatment will be defined as ((End date of treatment – Date of first dose of treatment) + 1).

Percent compliance is defined as (total number of puffs of study treatment taken across study days/total expected puffs taken across study days) across all days of a subject's dosing between start of study treatment and last day on study treatment) x 100. 4 puffs a day are expected, with 2 puffs on the final day of treatment.

Exposure to IP, number of puffs/inhalations of IP and % compliance will be summarized by treatment using the safety analysis set.

## 4.2.4 Analysis of FRI data

The primary analyses will be conducted using the ITT population. Similar methods will be used for the analysis of each of siVaw and siRaw.

The Day 15 value for each parameter in each period will be analysed using a linear mixed effect model. It is anticipated that the data will be logarithmically transformed prior to analysis. A multi-level model will be used to incorporate the repeated measurements from the lobes for each subject.

The model will include fixed effects for period, treatment, lobe and treatment by lobe interaction. The model will not include treatment sequence unless that term is determined to be important (p<0.10). Lobe will be included as a random effect, within each subject. Heterogeneity across lobes (within subject) will be modelled using an unstructured variance-covariance matrix, with independence assumed between subjects.

If this model fit fails to converge a compound symmetry covariance structure will be considered to model correlation across lobes from the same patient. If necessary, a per-visit

composite from across all lobes may be formed in order to conduct analyses at the subject rather than the lobe level. This would be based upon a sum across all available lobes for a subject, scaled for the number of evaluable lobes.

Estimates will be produced of the difference between treatments taken across all lobes. Where logarithmic transformations have been made, estimates will be exponentiated and treatment effects presented as ratios. Estimates and standard errors will be reported along with 2-sided 95% confidence intervals and p-values. The Kenward-Roger approximation for degrees of freedom and correction of downward bias in the standard error of fixed effect parameters will be used.

For the primary FRI endpoints only, line-plots will be produced displaying Day1 and Day 15 absolute values by treatment and sequence at the individual patient level using the mean of data from available single lobes for each patient.

For the primary endpoints only, the mITT population will be used to produce sensitivity analyses using only patients with data from both periods without important protocol deviations. Similar mixed models will be used. Should no patients require exclusion then these sensitivity analyses will not be required.

For the primary endpoints only, a further model will be produced which includes covariates for baseline. The model will include fixed effects for period, treatment, lobe and treatment by lobe interaction, subject-average baseline by lobe and period-dependent baseline by lobe. Both versions of baseline are continuous covariates. The use of both subject-average and period-dependent baselines allows for different coefficients for the between and within subject covariate regressions (Kenward and Roger 2010). Period-dependent baselines will be summarised for the primary endpoints.

Similar analyses to the primary analysis will be conducted for secondary and other efficacy endpoints based upon FRI, with the exception of the mass of deposited particles, the Internal Airflow Distribution and Air Trapping. For these values, only descriptive summaries will be produced by showing the deposition in each region of the patient's lungs at baseline. For the Internal Airflow Distribution, the presented values will consist of distance to normal values.

# 4.2.5 Spirometry / Body Plethysmography data

For spirometry and body plethysmography parameters data will be at the subject level and not split by lobe. The change from baseline to Day 15 for each endpoint will be analysed using a linear mixed effect model including subject-average baseline as a continuous covariate and treatment and period as fixed effects. The model will not include treatment sequence unless that term is determined to be important (p<0.10). The ITT population will be used. It is expected that plethysmography endpoints may require logarithmic transformation, but that spirometry endpoints will not.

# 4.2.6 Assumptions Checks and Removal of Outliers in Sensitivity Analyses

It is expected that logarithmic transformations will be required for most FRI and plethysmography endpoints, with the exception of the percent predicted lobe volume. Data

will be transformed via the natural logarithm prior to analysis and the adjusted mean estimates and confidence intervals from the linear models will be exponentiated back for presentation. As such the treatment effect for these endpoints will be presented as a ratio.

Under certain circumstances, (eg, during a COPD exacerbation unrelated to treatment) extreme and atypical values can arise. Such values may disproportionately affect model-based estimates of the fixed effect and variance parameters. Depending on the plots of the standardized residuals versus fitted values of the mixed-effect models, other data transformations may be considered. If necessary, this may include the fifth root, adapted for positive and negative values: fifthroot  $(x) = sign(x) * (abs(x)) ^ (1/5)$ .

For resistance measures, outliers can occur that are real values but affect the model estimates extremely. In these cases, values that are larger than the third quantile + 3 times the interquartile range may be removed. Infinite values for resistance are possible and these will be listed, but will be removed from the data before statistical analysis. If erroneous values are detected, every effort will be made to correct them prior to database lock. However, if these values cannot be corrected, they will be considered for removal from the analysis.

# 4.2.7 Exploratory analyses

In order to gain extra insights in the mode of action of the product, additional exploratory analyses may be executed and these may be reported outside of the CSR. These may entail post-hoc tests on the previously generated mixed-effect model. Contrasts for lobe by treatment interactions may be studied to examine the consistency of effects across the 5 lung lobes.

Pearson or Spearman's rank correlations between variables may be produced (depending upon behaviour of distributions). If appropriate, exploratory analyses of mixed-effect regressions or linear regression between parameters may be conducted to investigate associations between parameters, but these reported outside of the CSR.

## 4.2.8 Safety data

Adverse events will be summarized by the number and percentage of subjects experiencing an event. Tables will show the overall incidence of AEs, and the incidence for each treatment. Treatment emergent adverse events from the time of randomization onwards will be summarised. AEs reported as starting during a Washout Period or follow-up period will be assigned to the last treatment received.

AEs will be presented according to MedDRA preferred term and system organ class. Summaries will be produced by severity, seriousness, AEs leading to discontinuation, and by causality assessment to study drug. No hypothesis tests will be performed.

Clinically relevant findings from laboratory, ECG and vital sign parameters will be reported as adverse events. As such these assessments will not be further tabulated.

# 5. INTERIM ANALYSES (NOT APPLICABLE)

No interim analyses are planned in this study.

## 6. CHANGES OF ANALYSIS FROM PROTOCOL

The clinical study protocol stated that all FRI, spirometry and body plethysmography endpoints would utilise changes from baseline for statistical analyses. Effects were defined as differences between Day 15 and Day 1. As described in Kenward and Roger, conditioning on period-dependent baselines in a cross-over study has the potential to increase the variability of treatment effect estimates (Kenward and Roger 2010). For this reason statistical analyses will now be conducted either using absolute values or relative to subject-average (period independent) baselines.

It is now planned that FRI endpoints will be analysed using their absolute values at Day 15 rather than the change from baseline. This avoids the need to derive baselines across multiple lobes. In a cross-over study comparisons are driven by within-subject comparisons and the adjustment for baselines is not necessary as this adjusts for between patient variability.

Spirometry and plethysmography endpoints will utilise change from a subject-average baseline. The use of the subject-average baseline covariate will not affect the treatment effect estimates, but will allow for the estimation of changes from baseline for each separate treatment.

Given that the ITT, mITT and safety populations are expected to only differ slightly demographics and other characteristics will only be summarised for the ITT population. The mITT population will purely be used for sensitivity analyses of the primary endpoints should the ITT and mITT populations differ.

## 7. REFERENCES

R Core Team (2016). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL https://www.R-project.org/.

De Backer L, Vos W, De Backer J, Van Holsbeke C, Vinchurkar S, De Backer W. The acute effect of budesonide/formoterol in COPD: a multi-slice computed tomography and lung function study. Eur Respir J. 2012 Aug 1;40(2):298–305.

Kenward MG, Roger JH. The use of baseline covariates in crossover studies. Biostatistics (2010), 11, 1, 1–17

# 8. APPENDIX